CLINICAL TRIAL: NCT03891420
Title: A Phase 1b Double-blind, Placebo-controlled, Dose-ranging Study to Evaluate the Safety, Pharmacokinetics, and Anti-viral Effects of Galidesivir Administered Via Intravenous Infusion to Subjects With Yellow Fever or COVID-19
Brief Title: A Study to Evaluate the Safety, Pharmacokinetics and Antiviral Effects of Galidesivir in Yellow Fever or COVID-19
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor decision to no longer pursue indications studied in this trial
Sponsor: BioCryst Pharmaceuticals (Industry)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BCX4430-108; 272201300017C-18-0-1 (NIH); DMID18-0022 (Other: NIAID)
Record Dates: First submitted 2019-03-15; First posted 2019-03-27 (Actual); Last update posted 2021-05-27 (Actual); Status verified 2021-05

CONDITIONS: COVID-19; Yellow Fever
Keywords: COVID-19; Galidesivir; Yellow Fever
MeSH Terms: conditions — COVID-19; Yellow Fever | interventions — galidesivir

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Galidesivir (Experimental): Galidesivir IV infusion
  Interventions: Drug: Galidesivir
- Placebo (Placebo Comparator): Placebo IV infusion
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Galidesivir — Galidesivir IV infusion
  Arms: Galidesivir
Drug: Placebo — Placebo IV infusion
  Arms: Placebo

SUMMARY:
This is a placebo-controlled, randomized, double-blind study to evaluate the pharmacokinetics, safety and antiviral activity of galidesivir in subjects with yellow fever (YF) or COVID-19.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled study to evaluate the pharmacokinetics (PK), safety, and antiviral effects of galidesivir administered via intravenous (IV) infusion vs. placebo in hospitalized adult subjects with either Yellow Fever (Group A) or COVID-19 (Group B). The study will be conducted in two parts, and each Group (A or B) will proceed independently through the study. Part 1 is a dose ranging study with three sequential cohorts of eight patients each that will be randomized 3:1 to receive IV galidesivir or placebo every 12 hours for 7 days. Upon completion of part 1, an optimized dosing regimen of galidesivir will be selected for part 2, based on part 1 results including safety, PK, viral load reduction, and improvement in signs and symptoms and clinical manifestations, and mortality. In part 2, up to 42 patients will be randomized 2:1 to receive IV galidesivir or placebo. After treatment, the patients will remain hospitalized until resolution of symptoms allows release. All patients will be followed for mortality through Day 56.

ELIGIBILITY:
Inclusion Criteria: Group A - Yellow Fever

* Ability to provide written informed consent
* Males and nonpregnant, non-breast-feeding females, aged 18 years or older
* Subject weight ≥ 50 kg (110 lb.)
* Positive test for YFV by molecular amplification of the virus in the blood
* First onset of symptoms of YF occurring within the previous 7 days
* Male and female subjects must agree to the contraception requirements and must meet the inclusion criteria regarding contraception as outlined in the protocol
* CLCR of at least 60 mL/min by Cockcroft-Gault equation
* AST < 5000 u/L
* Indirect bilirubin < 1.5 mg/dL
* Neutrophil count < 7500 /mm3
* International Normalized Ratio (INR) < 1.5

Exclusion Criteria: Group A - Yellow Fever

* Any clinically significant medical condition or medical history that, in the opinion of the investigator or sponsor, would interfere with the subject's ability to participate in the study or increase the risk of participation for that subject
* Employment by the study site, or an immediate family relationship to either study site employees or Sponsor employee
* Lack of suitable veins for venipuncture/cannulation as assessed by the Investigator at Screening
* Participation in any other investigational drug or vaccine study currently or within the past 30 days
* Diagnosis of YF vaccine-related viscerotropic disease
* Subjects with hepatic encephalopathy as defined by Conn Score ≥ 1.
* Subject has severe immunosuppression or immunodeficiency, leukemia, lymphoma, thymic disease, generalized malignancy, or radiation therapy (within the past 3 months), or is undergoing current treatment with immunosuppressive drugs, defined as drugs that impair immune responses to infections
* A treatment plan for YF that would include concomitant administration of antiviral medications

Inclusion Criteria Group B - COVID-19

* Ability to provide written informed consent, accept randomization to any assigned treatment arm, and comply with planned study procedures
* Males and nonpregnant, non-breast-feeding females, aged 18 years or older
* Male and female subjects must agree to the contraception requirements and must meet the inclusion criteria regarding contraception as outlined in the protocol
* Subject weight ≥ 50 kg (110 lb.)
* Clinical syndrome consistent with moderate-severe (but not critically ill) COVID-19, defined by at least one of the following:

  1. Symptoms of acute viral lower respiratory tract infection, such as fever, non-productive cough, dyspnea, and either 1) a pulse oximetry oxygen saturation (SpO2) ≤ 94% or a respiratory rate > 24 breaths/minute as measured at rest without use of supplemental oxygen or 2) a clinical requirement for supplemental oxygen treatment or non-invasive mechanical ventilation
  2. Radiographic pulmonary findings seen on chest imaging (chest X-ray or computed tomography [CT scan]) consistent with COVID-19
* Positive test for SARS-CoV-2 by molecular amplification of the virus in a respiratory specimen (nasopharyngeal, oropharyngeal, lower respiratory tract [eg, expectorated sputum]) collected < 96 hours prior to randomization. Note: subjects may have a positive test recorded prior to screening if they are admitted to the hospital with a presumed case of COVID-19

Exclusion Criteria: Group B - COVID-19

* Any clinically significant medical condition or medical history that, in the opinion of the investigator or sponsor, would interfere with the subject's ability to participate in the study or increase the risk of participation for the subject
* Lack of suitable veins for venipuncture/cannulation as assessed by the Investigator at Screening
* Participation in any other investigational drug or vaccine study currently or within the past 30 days
* A clinical treatment plan that would include concomitant administration of any other experimental treatment or off-label use of marketed medications that are intended as specific treatment for the COVID-19 clinical syndrome or the SARS-CoV-2 infection. Any such medications must be discontinued prior to study enrollment, unless a formal written standard of care policy document from the national, state, or institutional authorities requires otherwise.
* Severe or rapidly progressive disease or medical condition of any type such that death is an expected or likely outcome within 72 hours or that would require referral or transfer to another medical facility
* Severe renal impairment (estimated glomerular filtration rate (eGFR) ≤ 50 mL/min/1.73m2) or receiving continuous renal replacement therapy, hemodialysis, or peritoneal dialysis
* Severe liver disease by medical history or ALT or AST > 5 times upper limit of normal
* Congestive heart failure by medical history ≥ Class 3
* Requiring invasive mechanical ventilation or extracorporeal membrane oxygenation (ECMO) at the time of randomization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2020-04-09 (Actual); Primary Completion 2021-01-31 (Actual); Study Completion 2021-04-30 (Actual)

PRIMARY OUTCOMES:
number of subjects with treatment emergent adverse events and serious adverse events | absolute number through the end of the study, approximately 56 days
number of subjects with change in laboratory parameters | absolute number and change from baseline through the end of the study, approximately 56 days
exposure of galidesivir as measured by plasma concentrations | 24 hours post dose on Day 1 through 12 hours post dose on Day 7

SECONDARY OUTCOMES:
yellow fever virus (YFV) titer (Group A) | change in YFV titer from baseline through Day 21
antiviral effect on SARS-CoV-2 in the respiratory tract - COVID-19 (Group B) | change in SARS-CoV-2 from baseline through Day 21
changes in clinical status using 8-point ordinal scale in COVID-19 (Group B) | through Day 21
changes from baseline and time to improvement using NEWS in COVID-19 (Group B) | through Day21
mortality | mortality at Day 56

CONTACTS AND LOCATIONS:
Overall Officials: Esper Kallas, MD, PhD, Principal Investigator — University of Sao Paulo, Brazil
Locations (5):
- Brazil (5):
  - Hospital de Clinicas da Universidade Federal do Parana, Curitiba, Paraná
  - Hospital Sao Vicente de Paulo-PPDS, Passo Fundo, Rio Grande do Sul
  - Hospital Sao Lucas da Pucrs, Porto Alegre, Rio Grande do Sul
  - Foundation Regional Faculty of Medicine of São José do Rio Preto, São José do Rio Preto, São Paulo
  - Clinical Research Unit and Department of Infectious and Parasitic Diseases Hospital das Clínicas, School of Medicine, USP, São Paulo, São Paulo

IPD SHARING:
Plan to Share IPD: No